CLINICAL TRIAL: NCT04426344
Title: Core Warming of COVID-19 Patients Undergoing Mechanical Ventilation: a Randomized, Single Center Pilot Study
Brief Title: Core Warming of COVID-19 Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal decision
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202005150
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: COVID 19
Keywords: COVID 19; Warming; Mechanical ventilation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized, single center pilot study
Who Masked: Participant
Masking Description: Due to the nature of this study, the physicians will not be blinded to the randomization assignment, however participants will be blinded. Once a subject is randomized, the research team will receive the randomization assignment (core warming or standard of care) and proceed with the procedures per the assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A - core warming (Experimental): Patients randomized to Group A will have core warming with the ensoETM device initiated in the ICU or other clinical environment in which they are being treated. The device will be used as indicated (for warming). Patient temperature measurement will be collected for both the core warming and standard of care arms during the study period (72 hours).
  Interventions: Device: ensoETM device
- Group B - Control Group (No Intervention): Group B is serving as the control group who will not have the ensoETM device used.Control group patients will be managed as per standard of care currently utilized in the ICU, which will include the use of other methods of temperature management as warranted. This would include warming with a forced air blanket only in hypothermic patients (core temperature < 36°C) or antipyretic therapy for febrile patients, as requested by the treating physician.

INTERVENTIONS:
Device: ensoETM device — Core warming will be performed using standard technique per instructions for use for the esophageal heat transfer device. The esophageal heat transfer device will be set to 42°C temperature after initial placement, and maintained at 42°C for the duration of treatment. It is expected that patient temperature will increase from baseline by 1°C to 2°C, but due to ongoing heat loss from the patient, the expected maximum patient temperature is below 39°C. The time course of illness of COVID-19 is such that most patients no longer have fever by the time of mechanical ventilation.[41] If patient temperature increases above this range and reaches 39.8°C, the device will be set to an operating temperature of 40°C, thereby preventing any further increase in patient temperature (ambient heat loss precludes patient from reaching device operating temperature).
  Arms: Group A - core warming

SUMMARY:
This is a small scale pilot study to evaluate if core warming improves respiratory physiology of mechanically ventilated patients with COVID-19, allowing earlier weaning from ventilation, and greater overall survival. This prospective, randomized study will include 20 patients diagnosed with COVID-19, and undergoing mechanical ventilation for the treatment of respiratory failure. Patients will be randomized in a 1:1 fashion with 10 patients (Group A) randomized to undergo core warming, and the other 10 patients (Group B) serving as the control group who will not have the ensoETM device used. Patients randomized to Group A will have core warming initiated in the ICU or other clinical environment in which they are being treated after enrollment and provision of informed consent from appropriate surrogate or legally authorized representative.

DETAILED DESCRIPTION:
Participants will be randomized in a 1:1 fashion to core warming with the study device (ensoETM) or to standard of care (standard temperature management and treatment). The device will be used as indicated (for warming). Patient temperature measurement will be collected for both the core warming and standard of care arms during the study period (72 hours).

Core warming will be performed using standard technique per instructions for use for the esophageal heat transfer device. The esophageal heat transfer device will be set to 42°C temperature after initial placement, and maintained at 42°C for the duration of treatment. It is expected that patient temperature will increase from baseline by 1°C to 2°C, but due to ongoing heat loss from the patient, the expected maximum patient temperature is below 39°C. The time course of illness of COVID-19 is such that most patients no longer have fever by the time of mechanical ventilation. If patient temperature increases above this range and reaches 39.8°C, the device will be set to an operating temperature of 40°C, thereby preventing any further increase in patient temperature (ambient heat loss precludes patient from reaching device operating temperature).

Control group patients will be managed as per standard of care currently utilized in the ICU, which will include the use of other methods of temperature management as warranted. This would include warming with a forced air blanket only in hypothermic patients (core temperature < 36°C) or antipyretic therapy for febrile patients, as requested by the treating physician. Episodes of hypothermia are infrequent and transient in this population, and the current standard of care generally utilizes a permissive approach to fever (allowing patients to remain mildly febrile) which will continue in the control group without modification (no intentional elevation of temperature will be provided in the control group).

Follow up data will be collected at 1 month following enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above the age of 18 years old.
2. Patients with a diagnosis of COVID-19 on mechanical ventilation.
3. Patient maximum baseline temperature (within previous 12 hours) < 38.3°C.
4. Patients must have a surrogate or legally authorized representative able to understand and critically review the informed consent form.

Exclusion Criteria:

1. Patients without surrogate or legally authorized representative able to provide informed consent.
2. Patients with contraindication to core warming using an esophageal core warming device.
3. Patients known to be pregnant.
4. Patients with <40 kg of body mass.
5. Patients with DNR status.
6. Patients with acute stroke, post-cardiac arrest, or multiple sclerosis.
7. Patients with history of esophageal disease
8. Patients with a baseline epinephrine dose greater than 0.6 mcg/kg/min
9. Patients with atrial fibrillation, atrial flutter, or other multifocal atrial tachycardia with a heart rate greater than 110 beats per minute.
10. Patients on 0.2 mcg/kg/min or more of norepinephrine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Viral load measured in tracheal aspirate 72 hours after initiation of core warming | 72 hours
  This endpoint will be compared between patients receiving core warming and those randomized to undergo standard care (standard temperature management, with or without antipyretics as needed) in order to determine an initial estimate of effect size and provide data from which to design adequately powered investigation and apply appropriate statistical testing.

SECONDARY OUTCOMES:
PaO2/FiO2 ratio 72 hours after initiation of core warming | 72 hours
Duration of mechanical ventilation | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Anne Drewry, MD, Principal Investigator — Washington Univeristy School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Bonfanti N, Gundert E, Drewry AM, Goff K, Bedimo R, Kulstad E. Core warming of coronavirus disease 2019 (COVID-19) patients undergoing mechanical ventilation-A protocol for a randomized controlled pilot study. PLoS One. 2020 Dec 1;15(12):e0243190. doi: 10.1371/journal.pone.0243190. eCollection 2020. PMID 33259540